CLINICAL TRIAL: NCT06507020
Title: Health Education for Preventing Falls in Older Adults Living in the Community: a Factorial Randomized Controlled Trial
Brief Title: Health Education for Preventing Falls in Older Adults Living in the Community
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Center for Disease Control and Prevention (Other Government)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: GZCDC-ECHR-2024P0116
Record Dates: First submitted 2024-06-27; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Accidental Falls; Older Adults

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Fall prevention knowledge education & Exercise education & Home hazard reduction education (Experimental): Fall Prevention Education:
  Form a health education group for the intervention subjects to learn about fall prevention. The project team will teach through talks, discussions, and shared experiences to boost their understanding and concepts on preventing falls.
  Exercise Education:
  In group settings, the project team will instruct participants on exercises to prevent falls, focusing on balance, leg strength, and endurance, and demonstrate the use of assistive tools.
  Home Hazard Reduction:
  Staff will visit homes to assess and guide on reducing fall risks, teaching participants to identify and suggest changes to home environment hazards.
  Interventions: Behavioral: Fall prevention knowledge education; Behavioral: Exercise education; Behavioral: Home hazard reduction education
- Fall prevention knowledge education & Exercise education (Experimental): The intervention in this arm consists of the following two components： Component 1: Fall prevention knowledge education To organise the study subjects in the intervention group to set up a falls prevention health education activity group, in which the project team will disseminate the knowledge and concepts of falls prevention through lectures, discussions, questions and answers, and sharing, so as to enhance the knowledge base required by the study subjects to prevent falls as well as to cultivate the relevant concepts.
  Component 2: Exercise education Using the group activities of the intervention group, through lectures, demonstrations, on-site exercises and practices, the project team taught the intervention group participants fall prevention exercise skills such as improvement of balance function, enhancement of lower limb muscle strength, endurance exercise, etc., and the use of fall prevention related assistive tools.
  Interventions: Behavioral: Fall prevention knowledge education; Behavioral: Exercise education
- Fall prevention knowledge education & Home hazard reduction education (Experimental): The intervention in this arm consists of the following two components： Component 1: Fall prevention knowledge education To organise the study subjects in the intervention group to set up a falls prevention health education activity group, in which the project team will disseminate the knowledge and concepts of falls prevention through lectures, discussions, questions and answers, and sharing, so as to enhance the knowledge base required by the study subjects to prevent falls as well as to cultivate the relevant concepts.
  Component 2: Home hazard reduction education Through the staff's in-home assessment and guidance, the project team instructed the study participants to assess the fall-related home environment risk factors and make recommendations for modifications.
  Interventions: Behavioral: Fall prevention knowledge education; Behavioral: Home hazard reduction education
- Exercise education & Home hazard reduction education (Experimental): The intervention in this arm consists of the following two components： Component 1: Exercise education Using the group activities of the intervention group, through lectures, demonstrations, on-site exercises and practices, the project team taught the intervention group participants fall prevention exercise skills such as improvement of balance function, enhancement of lower limb muscle strength, endurance exercise, etc., and the use of fall prevention related assistive tools.
  Component 2: Home hazard reduction education Through the staff's in-home assessment and guidance, the project team instructed the study participants to assess the fall-related home environment risk factors and make recommendations for modifications.
  Interventions: Behavioral: Exercise education; Behavioral: Home hazard reduction education
- Fall prevention knowledge education only (Experimental): Fall prevention knowledge education:
  To organise the study subjects in the intervention group to set up a falls prevention health education activity group, in which the project team will disseminate the knowledge and concepts of falls prevention through lectures, discussions, questions and answers, and sharing, so as to enhance the knowledge base required by the study subjects to prevent falls as well as to cultivate the relevant concepts.
  Interventions: Behavioral: Fall prevention knowledge education
- Exercise education only (Experimental): Exercise education:
  Using the group activities of the intervention group, through lectures, demonstrations, on-site exercises and practices, the project team taught the intervention group participants fall prevention exercise skills such as improvement of balance function, enhancement of lower limb muscle strength, endurance exercise, etc., and the use of fall prevention related assistive tools.
  Interventions: Behavioral: Fall prevention knowledge education
- Home hazard reduction education only (Experimental): Home hazard reduction education:
  Through the staff's in-home assessment and guidance, the project team instructed the study participants to assess the fall-related home environment risk factors and make recommendations for modifications.
  Interventions: Behavioral: Fall prevention knowledge education
- Care as usual (No Intervention)

INTERVENTIONS:
Behavioral: Fall prevention knowledge education — Frequency of Intervention: 4 sessions, 60 mins each, weeks 1, 3, 5, 8.
  Intervention format：group intervention, 12-15 participants in one group.
  Intervention content: Elderly fall risks, home safety improvements, community hazard identification, behavior modification.
  Intervention tools: digital teaching PPTs.
  Intervention deliverers: 2 members per community, one as leader for organizing health ed. activities (lectures, discussions, exercises, Q&A), the other as assistant for support and participant safety during exercises.
  Arms: Exercise education only; Fall prevention knowledge education & Exercise education; Fall prevention knowledge education & Exercise education & Home hazard reduction education; Fall prevention knowledge education & Home hazard reduction education; Fall prevention knowledge education only; Home hazard reduction education only
Behavioral: Exercise education — Frequency of intervention: 4 sessions Duration of intervention: 30 minutes/session, once in each of the 1st, 3rd, 5th and 8th weeks of the intervention period.
  Intervention format: group intervention, 12 people in a group (in principle, no more than 15 people).
  Intervention content: The content of health education included (1) basic knowledge of exercise safety, 4 methods of balance function exercise (2) review 4 methods of balance function exercise(3) methods of exercising muscle strength (4) 2 methods of endurance exercise.
  Intervention tools: accompanying teaching materials Intervention deliverers: same as before.
  Arms: Exercise education & Home hazard reduction education; Fall prevention knowledge education & Exercise education; Fall prevention knowledge education & Exercise education & Home hazard reduction education
Behavioral: Home hazard reduction education — Intervention Time:
  One home fall risk assessment and modification instruction at week 6 of health education.
  Frequency of Intervention:
  Single session.
  Intervention Format:
  Project staff conduct in-home fall risk assessments by appointment.
  Intervention Content:
  1. Evaluate fall risks in elderly living areas.
  2. Provide personal guidance, complete two written forms-one for records, one for the participants.
  3. Supply night lights, anti-slip mats, warning signs, and carpet mats; more services encouraged where possible.
  Intervention Tools:
  Utilize "Elderly Home Fall Risk and Retrofitting Guide" for detailed assessments and suggestions. Include tools like night lights, mats, and signs.
  Intervention Deliverers:
  Skilled community social workers or community health center staff.
  Arms: Exercise education & Home hazard reduction education; Fall prevention knowledge education & Exercise education & Home hazard reduction education; Fall prevention knowledge education & Home hazard reduction education

SUMMARY:
This clinical trial aims to evaluate the effectiveness of three health education intervention modules in preventing falls among older adults living in the community. The study is designed as a factorial randomized controlled trial, assessing the impact of three health education intervention modules: Fall prevention knowledge education，Exercise education, and Home hazard reduction education. Each module will have a 'yes' and 'no' version, resulting in eight experimental conditions.

The primary questions it seeks to address are: (1) What is the main effect of different health education intervention modules on preventing falls in older adults living in the community? (2)What is the interactive effect of different health education intervention modules on preventing falls in older adults living in the community?

The trial will be conducted in twenty four sub-district in Baiyun District, Guangzhou City. An estimated 37 participants will be recruited from each of the 24 sub-districts, with the sub-districts being randomly assigned to one of the eight experimental groups by a statistician independent of the research team using computer-generated random numbers.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 inclusive
* Live in the community
* Expected to live in their current place of residence for the next 12 months
* can walk 50 metres without the assistance of an assistive device

Exclusion Criteria:

* Exclusion of subjects with acute illness or acute stages of chronic disease

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 888 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of falling in each group | Baseline, 6-month, 12-month
  Falls will be monitored with supplied monthly fall diaries.

SECONDARY OUTCOMES:
Fall efficacy in each group | Baseline, 6-month, 12-month
  Fall efficacy will be monitored with 'Falls Efficacy Scale International, FES-I', and each item is scored on a scale of 1 to 4 (from "not at all confident" to "very confident"), with a total score of 16 to 64, with higher scores indicating a greater sense of fall efficacy or self-confidence.
Quality of life in each group | Baseline, 6-month, 12-month
  Quality of life will be monitored with 'the 12-item MOS Short-form Health Survey version 2, SF-12 V.2'. All entries except 1, 8, 9 and 10 are positively scored and the total score is calculated by the scale's unique standardised method, with a minimum score of 0 and a maximum score of 100

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT06507020/Prot_SAP_ICF_000.pdf